CLINICAL TRIAL: NCT03970863
Title: China Medical University Hospital, Taichung, Taiwan
Brief Title: Focal Therapy for Localized Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: difficulty in recruiting participants
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Po-Fan Hsieh, Attending Urologist, Department of Urology, China Medical University Hospital, China Medical University Hospital
Other Study IDs: CMUH107-REC3-119
Record Dates: First submitted 2019-05-27; First posted 2019-06-03 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Prostate Health Index — Use Prostate Health Index for the follow-up after focal therapy.

SUMMARY:
To evaluate the cancer control for prostate cancer patients treated with focal therapy.

DETAILED DESCRIPTION:
Traditional treatments for localized prostate cancer are radical prostatectomy and radiotherapy. However, they would carry side effects including urinary incontinence, sexual dysfunction, radiation cystitis and proctitis, leading to great impact on quality of life. Focal therapy of is another emerging treatment strategy for localized prostate cancer. It aims on ablation of the tumor with sparing of healthy prostatic tissue in order to minimize the injury to urinary and sexual function. Besides, owing to the improvement of multiparametric magnetic resonance imaging (mpMRI), the investigators can localize the prostate cancer more precisely and the accessibility of focal therapy is also increased.

Literature showed focal ablation of HIFU or cryotherapy for low and intermediate-risk prostate cancer patients yielded in brilliant outcomes. Biopsy in post-treatment one year showed 87% and 94.6% were negative for clinically significant cancer, respectively. Up to 92% of patients did not need salvage treatment in two years. Ninety-one to one hundred precent of patients had no urinary incontinence, and 74% and 81.5% had no erectile dysfunction, respectively.

This prospective study aims to evaluate the cancer control and quality of life for prostate cancer patients treated with focal therapy.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven unilateral prostate cancer, the other side insignificant cancer (Gleason 6 or less and maximal cancer core length 4mm or less) is allowed
* clinical T2a or less
* Gleason 4+3 or less
* serum PSA less than 20 ng/mL

Exclusion Criteria:

* T2b or higher
* Gleason 4+4 or higher
* serum PSA 20 or higher
* lymph node or distant metastasis
* previous treatment with prostatectomy, radiotherapy, androgen deprivation therapy, HIFU, or cryoablation

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostate cancer patients in a tertiary referral center in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-11-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
oncological outcome | 6 months
  MR/US fusion prostate biopsy to see if there is recurrent cancer
biochemical outcome | 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  change of Prostate Health Index (PSA, free PSA, and p2PSA will be combined to report PHI)

SECONDARY OUTCOMES:
Functional outcome | 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  change of Uroflowmetry, including maximal flow rate in milliliter per second and post-void residual volume in milliliter
Functional outcome | 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  change of IPSS questionnaire
Functional outcome | 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  change of OABSS questionnaire
Functional outcome | 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  change of IIEF-5 questionnaire
Functional outcome | 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  change of EORTC QLQ-30/PR-25 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Po-Fan Hsieh, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan